CLINICAL TRIAL: NCT06231654
Title: Use of Remote Photoplethysmography to Measure Heart Rate and Respiratory Rate in Pediatrics Compared to Standard Acquisition System: Prospective Comparative Trial
Brief Title: Evaluation of Remote Photoplethysmography to Assist Vital Signs Measure in Pediatrics
Acronym: rMonitoped1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-HNCL-06
Record Dates: First submitted 2023-12-21; First posted 2024-01-30 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Using Remote Photoplethysmography for Physiological Parameters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patents (Experimental): the child will be placed in a dedicated, quiet, well-lit office with their parents. The following data are then collected: sex, age, phototype according to Fitzpatrick's classification. The child sits in a chair facing a camera connected to a laptop running Caducy® Medical Device software. At the same time, and following the usual procedure, three ECG electrodes will be positioned on the patient.
  Interventions: Device: Remote photoplethysmography for physiological parameters

INTERVENTIONS:
Device: Remote photoplethysmography for physiological parameters — Patients participating in the study will be recruited from our emergency department.
  The child will be placed in a dedicated, quiet, well-lit office with their parents. The following data are then collected: sex, age, phototype according to Fitzpatrick's classification. The child sits in a chair facing a camera connected to a laptop running Caducy® Medical Device software. At the same time, and following the usual procedure, three ECG electrodes will be positioned on the patient. The whole device is connected to our standard device. Once the child is immobile and ready, the Caducy® application is launched. At the same time, our standard device is activated. After 30 seconds, we will collect the HR and FR values revealed by the Caducy® application via the non-contact plethysmography method. On the other hand, it will collect the HR and FR values revealed by our standard device (Mindray® scope).

SUMMARY:
Introduced in 1930, photoplethysmography techniques presented the possibility of measuring SpO2 and heart rates (HR) using the absorption of light by the blood to define these signals. In recent years, a new approach to photoplethysmography to measure physiological parameters without contact has been developed. This technique, called remote Photoplethysmography Imaging (rPPG), uses the different Red - Green - Blue color spectra at a skin captured by the camera video to determine a plethysmography signal. However, it has never been studied in pediatric patients. The objective is to evaluate the remote photoplethysmography technology to measure vital signs in pediatrics

DETAILED DESCRIPTION:
When assessing a child's clinical condition, the vulnerability of the child means is the needs to assess quickly and simply his vital status. Although several parameters are available to evaluate a potential life-threatening condition in pediatrics, the initial measurement of vital constants provides the clinician an immediate assessment about how much the vital status of the child is good or not. More particularly, heart rate (HR), respiratory rate (RR), oxygen saturation and blood pressure are defined as objective markers of a child's circulatory and respiratory status. In practice, manual measurements such as pulse palpation or thoracic ampliation counting are obsolete. A number of methods of measure are commonly used. Electrical recording via ECG electrodes or pulse counting via an oximeter can be used to measure heart rate. Respiratory rate can be measured using chest electrodes to assess its ampliation. In any emergency room, the collection of these constants requires a variety of medical devices that are usually time-consuming and human resources to collect them exhaustively and reliably. Moreover, these measurements may not be carried out under optimal conditions with children who may not be compliant, with as a result a lack of reliability or a missing measurement.

In adults, new and innovative measurement methods have emerged that offer acceptable reliability and accuracy compared with current reference methods. These include remote photo-plethysmography (rPPG), a process that enables vital constants to be assessed using a simple camera recording of the face over a short period of time.

Photoplethysmography (PPG) detect blood volume in the micro-vessels of tissues on the skin's surface. With each heartbeat, the volume in the arteries and arterioles changes. It is this variation that is measured using a LED placed mostly on the finger, ear or forehead.

Remote photoplethysmography (rPPG) is a non-invasive optical method for detecting pulse waves generated by the heart through measurements of peripheral blood perfusion. This technology may replace standard medical devices because of its ease of use, its low cost, its safety, convenience and its ability to offer multiple physiological assessments.

The company I-Virtual has enabled the development of this technique, whose technology is based on the analysis of different skin color spectra in the face, in order to determine a signal at the origin of these constants.

The Caducy® application using the rPPG technique can be downloaded onto a wide range of media. Using this app is quick and easy and requires to take a selfie using any camera available on a smartphone, tablet or computer at a sufficient distance ( the whole face should be visible on the screen). The application then takes between 30 seconds and 1 minute to analyze the various parameters. On January 25, 2023, i-Virtual obtained CE Class IIa certification for its Caducy® medical device, which measures vital signs via webcam. It thus became the first company in the world with this type of technology to obtain CE marking.

However, it has never been studied in pediatric patients. And yet, this easy-to-use, fast, material-saving application, certified for adult patients, could alleviate the difficulties of measuring vital signs in pediatrics that's mentioned earlier. In partnership with I-Virtual, the investigator would therefore like to test the use of remote photo-plethysmography or rPPG via its Caducy® application in pediatrics. The objective of the study is to evaluate the use of remote photoplethysmography to measure heart rate and respiratory rate in pediatric patients compared to standard acquisition system

ELIGIBILITY:
Inclusion Criteria:

* Children under 18 and over 3 years of age
* Any reason for consultation or hospitalization
* Written and signed informed consent from one parent or the person with parental authority,
* Membership of a social security scheme

Exclusion Criteria:

* Patient with a neurocognitive disorder
* Patient in immediate vital distress,
* Known cardiac arrhythmia,
* Scleroderma
* Patients suffering from pathological tremors or muscle spasms that prevent them from remaining static for the duration of the measurement.
* Parents who do not understand and/or speak French

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-07-02 (Estimated); Study Completion 2026-07-02 (Estimated)

PRIMARY OUTCOMES:
measure of heart rate (HR) with remote photo-plethysmography (rPPG) at 30 seconds of recording | at inclusion
  Assess the reliability of HR measurement using the rPPG at 30 seconds of recording versus that measured using ECG electrodes, the method taken as the gold standard, in a pediatric population

SECONDARY OUTCOMES:
HR measurement using rPPG at 60 seconds of recording | at inclusion
  Evaluate the reliability of HR measurement using rPPG (60-second recording) compared to ECG electrodes
RR measurement using rPPG (60-second recording) | at inclusion
  Evaluate the reliability of RR measurement using rPPG (60-second recording) compared to electrode system.
RR measurement using rPPG (30-second recording) | at inclusion
  Evaluate the reliability of RR measurement using rPPG (30-second recording) compared to electrode system.
RR measurement using rPPG according to the age ranges ranking | at inclusion
  Evaluate the reliability of RR measurement using rPPG at 30-second recording according to the age ranges ranking as the different periods of childhood [3y-7y[, [7y-12y[, [12y-18y[ and the patient phototype according to Fitzpatrick's classification
HR measurement using rPPG according to the age ranges ranking | at inclusion
  Evaluate the reliability of HR measurement using rPPG at 30-second recording according to the age ranges ranking as the different periods of childhood [3y-7y[, [7y-12y[, [12y-18y[ and the patient phototype according to Fitzpatrick's classification
parental satisfaction | at inclusion
  Evaluation of parental satisfaction with the application with likert Scale
failure rates of measurements | at inclusion
  Estimation of failure rates of measurements with each of the techniques (rPPG and electrodes).
Participant Satisfaction | at inclusion
  - Evaluation of participant satisfaction (children/adolescents aged 3-17 years) with the application with Likert Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Lenval - Hôpitaux Pédiatriques de Nice CHU-LENVAL, Nice, France

IPD SHARING:
Plan to Share IPD: No